CLINICAL TRIAL: NCT07084090
Title: Using IF-THEN Plans to Support Patients in Raising Safety Concerns About Their Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: University of Leeds (Other)
Responsible Party: Principal Investigator, Dr Chris Keyworth, Associate Professor, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025-22683-41374
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Patient Safety Concerns
Keywords: Patient safety; implementation intentions; behaviour change; safety concerns; randomised controlled trial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (volitional help sheet) (Experimental): Participants in this group will be asked to form implementation intentions-also known as "if-then" plans-specifically related to raising safety concerns. They will be presented with the stem: "If I am tempted not to raise concerns about my health care…" and provided with 10 evidence-based options to complete as many "if-then" plans as they wish. These options have been informed by behavioural science literature and have been shown to be effective in changing behaviours such as smoking cessation, reducing alcohol consumption, increasing physical activity, and reducing self-harm. Participants will link specific situations (the "if") with appropriate responses (the "then") using a structured online interface.
  Interventions: Behavioral: Implementation intention planning
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Implementation intention planning — Implementation intention planning to promote patient safety concerns
  Arms: Intervention (volitional help sheet)

SUMMARY:
The aim of the present research is to test the effectiveness of an implementation intention-based intervention for promoting the raising of safety concerns by patients in healthcare settings.

Each participant will be randomly allocated to one of two conditions: (1) a control condition, and (2) an intervention condition, in which participants form multiple implementation intentions (i.e. "if-then" plans) using a structured online interface. The main outcome measure will be the frequency with which participants report raising safety concerns in healthcare settings over a 12-month follow-up period.

DETAILED DESCRIPTION:
Background and study aims Previous research has demonstrated that while patients are often encouraged to raise concerns about the safety of their care, many feel uncertain about how and when to do so. This uncertainty can stem from a lack of confidence, fear of repercussions, or simply not knowing the appropriate channels. This study therefore aims to test whether a brief, theory-based intervention based on implementation intentions (Gollwitzer, 1993) can increase patients' confidence and likelihood of raising safety concerns in healthcare settings.

Implementation intentions, or "if-then" plans, are a well-established method for changing behaviour. They work by helping individuals identify critical situations ("if") and link them to specific responses ("then"), thereby automating helpful behaviours and overcoming barriers. This approach has been shown to be effective in changing a wide range of behaviours, including smoking cessation, reducing alcohol consumption, increasing physical activity, and reducing self-harm.

This study will examine whether forming "if-then" plans can help patients overcome barriers to raising safety concerns. The intervention will be delivered via an online questionnaire to a representative sample of adults in the United Kingdom, with follow-up after 12 months to assess changes in behaviour.

The aim of the study is to test the effectiveness of an implementation intention-based intervention for promoting the raising of safety concerns by patients in healthcare settings.

Aims To test the effectiveness of an implementation intention-based intervention for promoting the raising of safety concerns by patients in healthcare settings.

Who can participate? Adults aged 18 and over with good verbal and written understanding of English. Participants will be recruited from YouGov's existing panel of UK residents.

What does the study involve?

Participants will complete an online questionnaire about their experiences and attitudes toward raising safety concerns in healthcare. They will then be randomly assigned to one of two groups:

1. Intervention Group (Volitional Help Sheet with Implementation Intentions):

   Participants in this group will be asked to form implementation intentions-also known as "if-then" plans-specifically related to raising safety concerns. They will be presented with the stem: "If I am tempted not to raise concerns about my health care…" and provided with 10 evidence-based options to complete as many "if-then" plans as they wish. These options have been informed by behavioural science literature and have been shown to be effective in changing behaviours such as smoking cessation, reducing alcohol consumption, increasing physical activity, and reducing self-harm. Participants will link specific situations (the "if") with appropriate responses (the "then") using a structured online interface.
2. Control Group (Passive Control):

The (passive) control condition includes the same questionnaire as the experimental group, however participants are not presented with the intervention.

After 12 months, all participants will be invited to complete a follow-up questionnaire assessing how often they have raised safety concerns in healthcare settings.

What are the possible benefits and risks of participating? Participants may benefit by gaining confidence in raising concerns about their care. The study is low risk, and participants can withdraw at any time before data anonymisation. All data will be collected and stored securely by YouGov and anonymised before being shared with the research team.

Where is the study run from? The University of Manchester (United Kingdom) When is the study starting and how long is it expected to run for? July 2025 to May 2026 Who is funding the study? The NIHR Greater Manchester Patient Safety Research Collaboration (Greater Manchester Patient Safety Research Collaboration), at The University of Manchester.

Who is the main contact? Prof Christopher J. Armitage - chris.armitage@manchester.ac.uk Dr Chris Keyworth - c.keyworth@leeds.ac.uk

ELIGIBILITY:
Inclusion Criteria:

Aged 18 and over Good verbal and written understanding of English

Exclusion Criteria:

Aged under 18 years of age Poor verbal and written understanding of English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Raising safety concerns | 12 months
  Self-reported frequency of raising safety concerns at 12-month follow-up

SECONDARY OUTCOMES:
Capability, opportunity and motivation (based on COM-B model) | 12 months
  Measured using the Capability, Opportunity, Motivation questionnaire. Each of the items (0-10 scale) will be analysed separately as these each measure a separate construct. Higher scores indicate higher agreement with statements.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Keyworth C, Epton T, Goldthorpe J, Calam R, Armitage CJ. Acceptability, reliability, and validity of a brief measure of capabilities, opportunities, and motivations ("COM-B"). Br J Health Psychol. 2020 Sep;25(3):474-501. doi: 10.1111/bjhp.12417. Epub 2020 Apr 20. PMID 32314500
- [Result] Gollwitzer, P. M. (1993). Goal achievement: The role of intentions. European review of social psychology, 4(1), 141-185.